CLINICAL TRIAL: NCT04880395
Title: Dolutegravir-Lamivudine for naïve HIV-Infected Patients With ≤200 CD4/mm3
Acronym: DOLCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: ViiV Healthcare (Industry); Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Maria Ines Figueroa, MD, Fundación Huésped
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH 57
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
Keywords: antiretroviral naive triple therapy. Dolutegravir-Lamivudine; dual-therapy
MeSH Terms: interventions — Lamivudine; dolutegravir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : Dolutegravir plus Lamivudine (Experimental): DOVATO: Dolutegravir 50mg/lamivudine 300 mg, FDC, 1 coformulated tablet QD
  Interventions: Drug: Intervention Arm: dolutegravir/lamivudine
- active comparator : TDF/XTC plus Dolutegravir (XTC stands for lamivudine OR emtricitabine) (Active Comparator): Unit Dose:
  * TDF/FTC 300/200 mg, 1 coformulated tablet QD (FDC) plus Dolutegravir 50 mg, 1 tablet QD OR
  * TDF/3TC 300/300 mg, 1 coformulated tablet QD (FDC) plus Dolutegravir 50 mg, 1 tablet QD
  Interventions: Drug: Comparator ARM: TDF/XTC plus Dolutegravir (XTC stand for lamivudine OR emtricitabine)

INTERVENTIONS:
Drug: Intervention Arm: dolutegravir/lamivudine — 1 pill QD
  Other Names: Dovato
  Arms: Experimental : Dolutegravir plus Lamivudine
Drug: Comparator ARM: TDF/XTC plus Dolutegravir (XTC stand for lamivudine OR emtricitabine) — 1 pill of each QD
  Arms: active comparator : TDF/XTC plus Dolutegravir (XTC stands for lamivudine OR emtricitabine)

SUMMARY:
Protocol Title: DOLCE: Dolutegravir-Lamivudine for naïve HIV-Infected Patients with ≤200 CD4/mm3

Protocol Number: FH-57

Study Objectives: To assess the antiviral activity at week 48 of DTG+3TC among naïve HIV patients with a CD4 count ≤200 cells /mm3.

DETAILED DESCRIPTION:
Primary endpoint: Proportion of patients with viral load < 50 copies/mL at week 48 using the ITT-exposed analysis (FDA snapshot) for the intent-to-treat exposed (ITT-E) population.

Secondary Objectives:

* To assess the antiviral activity of DTG+3TC and DTG+TDF/XTC at week 24
* To evaluate the safety and tolerability of DTG+3TC and DTG+TDF/XTC over time
* To assess the antiviral activity of DTG+3TC and DTG+TDF/XTC at week 48 in patients with baseline viral load >100,000 c/mL
* To evaluate immunological activity (CD4+ lymphocyte [CD4 counts]) at Week 24 and Week 48
* To assess the development of HIV-1 resistance in patients with virologic failure or viral rebound treated with DTG+3TC or DTG+TDF/XTC
* To evaluate the incidence of disease progression (HIV-associated conditions, AIDS and death) of DTG + 3TC and DTG + TDF/XTC over time.

Secondary endpoints:

* Proportion of patients treated with DTG+3TC and DTG+TDF/XTC with HIV-1 levels of less than 50 copies/mL at week 24
* Frequency, type and severity of adverse events and laboratory abnormalities and proportion of patients who discontinue DTG+3TC or DTG+TDF/XTC due to adverse events or death
* Proportion of patients with baseline HIV-1 RNA >100,000 c/mL that achieve virological suppression at week 48 weeks,
* Changes in CD4 count, CD8 count and CD4/CD8 ratio between baseline and 48 weeks
* Number and type of resistance mutations in case of virologic failure (defined as a confirmed viral above 200 copies/mL after week 24 copies/mL or viral rebound at any timepoint)
* Incidence of IRIS and disease progression (HIV associated conditions, AIDS and death).

Tertiary objectives:

● TDF/XTCTo explore change in health-related quality-of-life for subjects treated with DTG plus 3TC and DTG + TDF/XTC

Tertiary endpoints:

● Change from Baseline in health-related quality of life using EQ-5D-5L and PHQ9 at Weeks 24, and 48

Patient Population:

HIV-1-infected subjects aged >18 years who are naïve to antiretroviral therapy with ≤200 CD4 cell/mm3

Study Design:

Prospective, Phase IV, randomized, multicenter, parallel group study design

Regimens:

Dolutegravir 50 mg /lamivudine 300 mg QD FDC. Dolutegravir 50 mg QD plus tenofovir 300 mg/emtricitabine 200mg or plus tenofovir 300 mg/ lamivudine 300 mg.

Duration: 48 weeks

Sample size:230 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB) / Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions.
2. Documented HIV-1 infection defined as a positive rapid test or ELISA plus a plasma HIV-1 RNA (>1,000 copies/mL) or a positive western blot. A previous result performed on the last 30 days can be used.
3. ≥18 years of age
4. Naïve to ARV therapies (defined as ≤ 10 days of prior therapy with any antiretroviral therapy following an HIV diagnosis). Previous use of PrEP or PEP is allowed if there is documented HIV seronegativity between the last prophylactic dose and the date of HIV diagnosis.
5. HIV RNA at screening visit > or = 1,000 copies/mL. A previous result performed on the last 30 days can be used.
6. CD4 at screening < or = 200 cells/mL A previous result performed on the last 30 days can be used.
7. Subjects can comply with protocol requirements.
8. Subject agrees not to take any medication during the study, including over-the-counter medicines or herbal preparations, without the approval of the trial physician.
9. Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the study.
10. A female may be eligible to enter and participate in the study if she is not pregnant (as confirmed by serum pregnancy test negative at screening, and a urine negative test at baseline), not lactating and at least one of the following condition applies:

    1. Women with non-reproductive potential, defined as pre-menospausal females with documented tubal ligation or hysterectomy, or bilateral oophorectomy; or as post-menospausal women defined as 12 months of spontaneous amenorrhea, and ≥45 years of age in women without hormonal replacement therapy.
    2. Women with reproductive potential and agrees to follow one of the contraceptive options listed in the Appendix 3 from at least 15 days prior to the first dose of medication and until at least 30 days after the last dose of study medication and completion of the follow-up visit.

Any contraception method must be used consistently, in accordance with the approved product label. All subjects participating in the study should be counselled on safer sexual practices including the use of effective barrier methods and the choice of effective contraceptive method should be documented in the eCRF.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or women who plan to become pregnant in the next year.
2. Subjects testing positive for Hepatitis B surface antigen (+HBsAg) at screening, or anticipated need for Hepatitis C virus (HCV) therapy with drugs with potential drug-drug interaction during the study.
3. Subjects with severe hepatic impairment (Child-Pugh class C), or unstable liver disease (ascites, encephalopathy, coagulopathy, or oesophageal or gastric varices) or cirrhosis.
4. Opportunistic infections that impede to start ART immediately (specifically tuberculosis, meningeal tuberculosis or cryptococcosis within the first month of specific treatment). Subjects with other suspected or confirmed active opportunistic infections and subjects with cryptococcal disease after the initial period can be included if she/he can follow the protocol and if her/his participation could benefit the subject. A clear documentation of these aspects must to be done in the clinical chart of the participant.
5. Subjects who in the investigator's judgment, pose a significant suicidality risk.
6. History or presence of allergy to the study drugs or their components or drugs of their class
7. Treatment with any of the following agents within 28 days of screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses; or treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening; or exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product.
8. Any previous evidence of resistance to dolutegravir (defined as the presence of G118R, Q148 H/K/R or R263K), to lamivudine (presence of the mutation M184V) or resistance to tenofovir (mutation K65R or more than 3 TAMs) with a Sanger sequence method or using next-generation sequencing (NGS) at a frequency >15%. If the subject does not have a previous resistance test, samples will be taken at the screening visit and the subject can be randomized and start the study. while awaiting the results (see section 4.8).
9. Any verified Grade 4 abnormality.
10. Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal (ULN), or ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin).
11. Creatinine clearance of <50mL/min via Cockroft-Gault method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ines Figueroa, PI, Principal Investigator — Fundación Huésped
Locations (11):
- Argentina (5):
  - Fundación Huésped, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital General de Agudos Dr. Cosme Argerich, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital de Infecciosas Francisco Javier Muñiz, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto CAICI, Rosario, Santa Fe Province
  - Hospital de Agudos J.A.Fernandez, Buenos Aires
- Brazil (6):
  - Fundação Bahiana de Infectologia, Salvador, Estado de Bahia
  - HUOC - Hospital Universitário Oswal do Cruz - Universidade de Pernambuco, Recife, Pernambuco
  - Hospital Geral de Nova Iguaçu, Nova Iguaçu, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa: Instituto de Infectologia Emílio Ribas, Pacaembu, São Paulo
  - Centro de Treinamento e Referência DST/AIDS, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
IPD available upon request. The request should be supported with a hypothesis-driven project, that should include analysis plan
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 month after last patient last visit
Access Criteria: By request

REFERENCES:
- [Derived] Figueroa MI, Brites C, Cecchini D, Ramalho A, Francos JL, Lacerda M, Rolon MJ, Madruga JV, Sprinz E, Souza TNL, Parenti P, Converso D, Mernies G, Sued O, Cahn P; DOLCE study group. Efficacy and Safety of Dual Therapy With Dolutegravir/Lamivudine in Treatment-naive Persons With CD4 Counts <200/mm3: 48-Week Results of the DOLCE Study. Clin Infect Dis. 2025 Aug 28:ciaf415. doi: 10.1093/cid/ciaf415. Online ahead of print. PMID 40874763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 17th, 2021 - May 04th, 2023. Sites from Argentina and Brazil.
Pre-assignment Details: Eligible participants were non-pregnant, not breastfeeding adults (18 years or older) living with HIV-1, ART naïve, having plasma HIV-1 (pVL) RNA ≥1,000 copies/mL and, CD4 cll counts≤ 200 cells/mm³ at screening. Key exclusión criteria included a positive Hepatitis B coinfection, pre-existing major viral resistance mutations to DTG, 3TC, or TDF, active opportunistic infections, liver or kidney disease.
Period: Overall Study
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Started | 153 (Two participants who were randomized to the active comparator arm received DTC/3TC by mistake and were considered as in the experimental arm for all the analyses. In addition, one participant randomized to experimental group was withdrawn before receiving any dose and therefore excluded from all analyses.) | 77
Completed | 140 | 71
Not Completed | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine) | Total
Number analyzed (Participants) | 153 | 77 | 230
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [29 to 48] | 34 [28 to 47] | 35 [28 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 21 | 56
  Male | 118 | 56 | 174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 26 | 9 | 35
  Race: Native | 8 | 0 | 8
  Race: White | 52 | 37 | 89
  Race: Other (Hispanic- Latino/Mixed) | 67 | 31 | 98
CD4 cell count [Median (Inter-Quartile Range); unit: cell/mL] | 109 [48.8 to 177] | 128 [58.5 to 200] | 116 [53.3 to 188]

OUTCOME MEASURES:

1. Primary Outcome: Antiviral Activity at Week 48 of DTG+3TC Among ART-naïve HIV Patients With a CD4 Count ≤200 Cells/mm3.
Description: Percentage of patients with viral load < 50 copies/mL at week 48 using the ITT-exposed analysis (FDA snapshot) for the intent-to-treat exposed (ITT-E) population.
Time Frame: Week 48
Population: One participant randomized to experimental arm was withdrawn before receiving any dose and therefore excluded from all analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 152 | 77
Participants | 125 | 62

2. Secondary Outcome: Antiviral Activity of DTG+3TC and DTG+TDF/XTC (TDF/FTC or TDF/3TC) at Week 24
Description: Percentage of patients treated with DTG+3TC and DTG+TDF/XTC with HIV-1 levels of less than 50 copies/mL at week 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 152 | 77
Participants | 110 | 58

3. Secondary Outcome: Safety and Tolerability of DTG+3TC and DTG+TDF/XTC Over Time
Description: Percentage of patients who discontinue treatment due to adverse events or death
Time Frame: week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 152 | 77
Participants | 7 | 2

4. Secondary Outcome: Antiviral Activity of DTG+3TC and DTG+TDF/XTC at Week 48 in Patients With Baseline Viral Load >100,000 c/mL
Description: Percentage of patients with baseline viral load >100,000 c/mL that reach HIV-1 levels of less than 50 copies/mL at week 48
Time Frame: Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 94 | 47
Participants | 76 | 36

5. Secondary Outcome: Changes in Lymphocytes Subsets Between Baseline and 48 Weeks
Description: Changes in lymphocytes CD4 cells count per mL
Time Frame: Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cell/mL
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 152 | 77
cell/mL | 200 [127 to 316] | 177 [128 to 267]

6. Secondary Outcome: Development of HIV-1 Resistance in Patients With Virologic Failure or Viral Rebound Whilst Being Treated With DTG+3TC or DTG+TDF/XTC
Description: Number and type of resistance mutations in case of virologic failure (defined as a confirmed viral above 200 copies/mL on or after week 24 or confirmed viral rebound at any timepoint)
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 18 | 9
Participants | 0 | 0

7. Secondary Outcome: Incidence of IRIS or Disease Progression (HIV Associated Conditions, AIDS and Death).
Description: Evaluation of disease progression incidence (HIV-associated conditions, AIDS and death) with DTG+3TC and DTG + TDF/XTC treatment over time
Time Frame: week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
Number analyzed (Participants) | 152 | 77
Participants | 9 | 6

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- Experimental : Dolutegravir Plus Lamivudine: Dolutegravir 50 mg/lamivudine 300 mg, FDC, 1 coformulated tablet QD
- Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine): * TDF/FTC 300/200 mg, 1 coformulated tablet QD (FDC) plus Dolutegravir 50 mg, 1 tablet QD, OR
  * TDF/3TC 300/300 mg, 1 coformulated tablet QD (FDC) plus Dolutegravir 50 mg, 1 tablet QD
  Data related to the use of TDF/3TC or TDF/FTC was not discriminated. Both options used were considered as a single treatment arm: TDF/XTC plus dolutegravir.
Arm/Group | Experimental : Dolutegravir Plus Lamivudine | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine)
All-Cause Mortality (participants affected / at risk) | 4/152 | 2/77
Serious Adverse Events (participants affected / at risk) | 15/152 | 9/77
Other Adverse Events (participants affected / at risk) | 37/152 | 21/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental : Dolutegravir Plus Lamivudine (N=152) | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine) (N=77)
Tuberculosis meningoencephalitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
IRIS in tuberculous meningitis (Nervous system disorders) | 1 (1) | 0 (0)
Possible lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bilateral herpetic retinitis (Eye disorders) | 0 (0) | 1 (1)
Burkitt's lymphoma (non-Hodgkin's lymphoma) (Immune system disorders) | 1 (1) | 0 (0)
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Probable aortic aneurysm rupture (Cardiac disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lymphoproliferative disorder with metástasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Ureteral rupture (Renal and urinary disorders) | 1 (1) | 0 (0)
Disseminated TB with meningeal involvement (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis and vitritis (Eye disorders) | 1 (1) | 0 (0)
Car accident (General disorders) | 0 (0) | 1 (1)
Hospitalization for investigation of pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Investigation of fever, disorientation and weight loss (Immune system disorders) | 0 (0) | 1 (1)
Esophagus substenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal tubular acidosis + Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pancytopenia febrile (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Probable pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Neurotoxoplasmosis (Nervous system disorders) | 0 (0) | 1 (1)
Cryptosporidiosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental : Dolutegravir Plus Lamivudine (N=152) | Active Comparator : TDF/XTC Plus Dolutegravir (XTC Stands for Lamivudine OR Emtricitabine) (N=77)
Insomnia/Nightmares (General disorders) | 6 (6) | 3 (3)
Itching/Rash/Prurigo (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Depressive symptoms/Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Abdominal pain/Epigastralgia/Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Weight gain (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Elevated transaminases (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hiperglucemia (Endocrine disorders) | 1 (1) | 1 (1)
Amylase elevation (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Creatinine increase (Renal and urinary disorders) | 1 (1) | 1 (1)
Malassezia folliculitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypercholesterolemia/ Dyslipidemia (Endocrine disorders) | 1 (1) | 0 (0)
Plateletopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
IRIS in Tuberculous meningitis (Nervous system disorders) | 1 (1) | 0 (0)
Disseminated Tuberculosis with meningeal involvement (Nervous system disorders) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pharmacodermia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cytomegalovirus retinitis (Eye disorders) | 0 (0) | 1 (1)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bilateral cervical lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Pancytopenia febrile (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Fever, diarrhea, abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lipid increase (Hepatobiliary disorders) | 1 (1) | 0 (0)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Ulcer in the left ear (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Glutamic Oxaloacetic Transaminase increase (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any documents, reports or data received or generated by PIs under the Agreement, including in particular those containing or reflecting specific information or the Study's results or data, may not be used, disclosed, communicated or published by PIs, whether for its own benefit or that of third parties, free of charge or against payment, in any country, without first obtaining the prior written permission of Fundación Huésped (Sponsor) in each instance.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04880395/Prot_SAP_000.pdf